CLINICAL TRIAL: NCT06809647
Title: A Prospective Interventional Cohort Study to Evaluate the Efficacy and Safety of the AquaLumen, a Novel Filtration Procedure for the Treatment of Open Angle Glaucoma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: PLU Ophthalmic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PLU-01
Record Dates: First submitted 2025-01-30; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Glaucoma Open-Angle
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- This is the group that will undergo the surgical treatment (Experimental)
  Interventions: Device: Glaucoma surgery

INTERVENTIONS:
Device: Glaucoma surgery — This is an implant-free, minimally invasive glaucoma surgery

SUMMARY:
The study will follow a group of patients with glaucoma disease that undergo a surgical procedure intended to reduce the intra-ocular pressure (IOP) for a period of one year.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe open angle glaucoma
* Central corneal thickness between 480 and 610 microns

Exclusion Criteria:

* surgical history of corneal graft
* presence of corneal opacities
* Failed prior trabeculectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-03-30 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Intra Ocular pressure | 12 months
Use of concomitant topical glaucoma medications | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- MUSC Storm Eye Institute, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided